CLINICAL TRIAL: NCT06723379
Title: A Genetic Survey of Cytochrome P450 2D6 Genotypes by Nanopore DNA Sequencing and Clinical Response to Codeine and Tramadol in Postoperative Pain Management
Brief Title: Genetics of Cytochrome CYP2D6 and Effects of Codeine and Tramadol on Postoperative Pain Management
Acronym: CYP2D6
Status: Completed | Type: Observational
Sponsor: Fraser Health (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Perseus Missirlis, Clinical Instructor, Fraser Health
Other Study IDs: 21-01422
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A single EDTA tube of 2-3 mL of blood will be collected in the OR as per standard procedure and the tube will be labelled in the standard way with a computer generated label containing the standard patient identifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy surgical patients: Healthy surgical patients who are undergoing surgical procedures with projected moderate postoperative pain.

SUMMARY:
Codeine is one of the most commonly prescribed opioids in the world. The speed at which our liver metabolizes codeine into morphine depends on an important protein called cytochrome P450 2D6 (CYP2D6). Many people across the world have different CYP2D6 metabolizing speeds. Codeine provides inadequate pain management to those who have slow-metabolizing CYP2D6. In contrast, codeine can be life-threatening to those who have rapidly-metabolizing CYP2D6 because of the abruptly high dose of morphine. By analyzing specific genes, we are able to predict a patient's response to medication, thus drug type and dosing can be tailored according to their genetics. The purpose of this study is to observe if nanopore CYP2D6 DNA genetic sequencing can classify patients according to their CYP2D6 phenotype and thus predict their response to codeine and tramadol. The overall project is to determine the practicality of a genetic survey of CYP2D6 for healthy patients undergoing surgical procedures.

DETAILED DESCRIPTION:
PURPOSE: The purpose of this study is to investigate if genetic variants of CYP2D6 are a predictive factor for postoperative pain management with conventional codeine and tramadol pain therapy. With CYP2D6 DNA analysis, we hope to be able to correlate a patients' genetics and their physiological response to conventional codeine and tramadol dosing.

RESEARCH QUESTION: Is CYP2D6 metabolizer status a predictive factor for the effectiveness of postoperative pain management with conventional pain therapy doses of codeine and tramadol?

HYPOTHESIS: Our hypothesis is that patients with known rapid metabolizing CYP2D6 variants will have higher incidences of opioid side effects with conventional opioid dosing. On the other hand, patients with known poor-metabolizing CYP2D6 variants will have inadequate pain management with conventional opioid dosing.

JUSTIFICATION: Understanding the relationship between CYP2D6 variants and conventional opioid dosing in a clinical setting will facilitate future studies that investigate personalized dosing in order to improve pain management and reduce risk of opioid side effects.

OBJECTIVES: The primary objective of this study is to determine the practicality of undertaking a medium-scale genetic survey of CYP2D6 for healthy patients undergoing surgical procedures. Secondary objectives include: investigate the feasibility of characterizing CYP2D6 genetic variants into one of four metabolizer groups, investigate if there is a distinguishable pattern between CYP2D6 metabolizer status and postoperative pain management quality with conventional pain therapy dosages such as codeine and tramadol, investigate if there is a distinguishable pattern between CYP2D6 metabolizer status and the presence of opioid side effects with conventional pain therapy dosages such as codeine and tramadol, to raise awareness of the clinical relevance of CYP2D6 variants on codeine and tramadol metabolism as well as the complications that arise from conventional, non-personalized pain management.

RESEARCH DESIGN: Prospective observational feasibility study of healthy elective surgical patients. Projected enrolment up to 50 participants. All participants receive standardized anesthetic with weight based dosing of opiates. Data collected will include: 2-3 ml blood sample taken prior to surgery under general anesthesia, DNA sequencing and genotype identification, chart review during post-operative care unit stay (PACU), and a survey administered by phone 24 after discharge from the PACU.

STATISTICAL ANALYSIS: Given the exploratory nature of this feasibility study and small convenience sample size, data will be summarized using descriptive statistics for most outcome variables. If possible, nonparametric statistical tests may be performed to look at associations between genetic variant and outcomes and differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 year and otherwise healthy (ASA 1 or 2)
2. Undergoing an elective outpatient surgical procedure at Royal Columbian Hospital or Eagle Ridge Hospital with projected moderate post-operative pain
3. Surgical procedure that requires general anaesthetic and post-operative pain management routinely managed with either codeine or tramadol by attending surgeon (i.e., ACL repair)
4. Attending surgeon routinely prescribes either tramadol or codeine for post-operative pain management

Exclusion Criteria:

1. Pre-existing chronic pain condition
2. Any psychiatric diagnosis, such as depression or anxiety (Lautenbacher et al., 1994)
3. History of substance abuse/dependence
4. Multiple medical comorbidities (a single well-controlled medical comorbidity will not be a contraindication - i.e., controlled hypothyroidism)
5. Allergy, sensitivity, or other contraindication to either codeine or tramadol
6. Regional anesthetic (inclusive either of a major peripheral nerve block or neuraxial anesthetic) planned by attending anesthesiologist)
7. Unable to provide informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For the pilot study, healthy patients (ASA 1 or 2) who are undergoing surgical procedures at Royal Columbian Hospital or Eagle Ridge Hospital with projected moderate postoperative pain will be selected. It is estimated that five patients will be approached to learn more about the study each week and 50-60% will consent to participate given the minimally invasive study procedures and the potential for participants to learn valuable personal pain medication metabolizing genetic status. Therefore, this study aims to enroll approximately ten patients per month up to a maximum of fifty total patients over a five-month span.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
CYP2D6 genotypes/phenotypes | 6 months
  CYP2D6 genotype determined by nanopore DNA sequencing which will be cross-referenced with published genotypes to determine CYP2D6 phenotype

SECONDARY OUTCOMES:
Total opiate consumption | 6 months
  Total opiate consumption (morphine milligram equivalents, continuous) observed immediately post-op, before tramadol or codeine administration, and 1 hour or later post tramadol/codeine administration
Pain scores | 6 months
  Pain scores (0 - 10, ordinal) observed immediately post-op, before tramadol or codeine administration, and 1 hour or later post tramadol/codeine administration
Sedation level | 6 months
  Sedation assessments (1 - 4, ordinal) observed immediately post-op, before tramadol or codeine administration, and 1 hour or later post tramadol/codeine administration
Administration of anti-nausea medications | 6 months
  Administration of anti-nausea medications (Yes/No, dichotomous) observed immediately post-op, before tramadol or codeine administration, and 1 hour or later post tramadol/codeine administration
Postoperative Day 1 current pain and worst pain since discharge | 6 months
  Current pain and worst pain since discharge (0 - 10, ordinal) at 24-hour post-op discharge telephone follow-up call
Postoperative Day 1 Nausea and vomiting (Yes/No, dichotomous) | 6 months
  Nausea and vomiting (Yes/No, dichotomous) at 24-hour post-op discharge telephone follow-up call.
Total opioids taken since discharge | 6 months
  Total opioids taken since discharge (morphine milligram equivalents, continuous) at 24-hour post-op discharge telephone follow-up call.

CONTACTS AND LOCATIONS:
Overall Officials: Perseus Missirlis, MSc, MD, Principal Investigator — Fraser Health
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No